CLINICAL TRIAL: NCT01406106
Title: EFFECT OF PLANT STEROLS ON THE LIPID PROFILE OF PATIENTS WITH HYPERCHOLESTEROLAEMIA. RANDOMISED, EXPERIMENTAL STUDY
Brief Title: Effect of Plant Sterols on the Lipid Profile of Patients With Hypercholesterolaemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gerencia de Atención Primaria, Albacete (Other)
Collaborators: Fundación para la Investigación Sanitaria en Castilla-La Mancha (FISCAM) (Unknown); Castilla-La Mancha Health Research Foundation. (Unknown)
Responsible Party: Ignacio Párraga Martínez, Gerencia de Atención Primaria de Albacete
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009/001
Record Dates: First submitted 2011-07-28; First posted 2011-07-29 (Estimated); Last update posted 2011-07-29 (Estimated); Status verified 2011-07

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; Lipids; Cardiovascular disease; Risks factors; Primary Care
MeSH Terms: conditions — Hypercholesterolemia; Cardiovascular Diseases | interventions — plant stanol ester

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liquid yoghurt with plant stanol esters (Experimental): Dairy product in the form of liquid yoghurt, marketed in Spain, that contains 2 g per container of plant stanol esters: sitostanol and campestanol (AHA recommended dose - 1.5 to 3 g).
  It also contains: proteins 1.8 g, carbohydrates 9.8 g, fat 1.4 g, plant stanol 2 g, vitamin B6 0.6 mg, folic acid 60 mg.
  Interventions: Dietary Supplement: Plant stanol esters
- Yoghurt without plant stanol esters (Placebo Comparator): Composition per container: proteins 1.8 g, carbohydrates 9.8 g, fat (except stanol) 1.4 g, plant stanol 2 g, vitamin B6 0.6 mg, folic acid 60 mg.
  Interventions: Dietary Supplement: Plant stanol esters

INTERVENTIONS:
Dietary Supplement: Plant stanol esters — The administration of a dairy product in the form of liquid yoghurt, marketed in Spain, that contains 2 g per container of plant stanol esters: sitostanol and campestanol (AHA recommended dose - 1.5 to 3 g). The enriched product and the placebo will have the same characteristics (composition and outward appearance), but the placebo will not contain stanol esters. The dose will be one container a day, after the main meal, for 24 months. The participants may continue with their previously prescribed lipid-lowering treatment and new treatment needed for this disease or for other diseases. Composition per container: proteins 1.8 g, carbohydrates 9.8 g, fat (except stanol) 1.4 g, plant stanol 2 g, vitamin B6 0.6 mg, folic acid 60 mg. The control group will receive one unit a day of yoghurt not supplemented with stanol esters that has a similar appearance to the enriched yoghurt.

SUMMARY:
Background information Studies have been conducted on supplementing the daily diet with plant sterol ester-enriched milk derivatives in order to reduce LDL-cholesterol levels and, consequently, cardiovascular risk. However, clinical practice guidelines on hypercholesterolaemia state that there is not sufficient evidence to recommend their use in subjects with hypercholesterolaemia. The null hypothesis establishes that there is no relationship between the decrease in blood LDL-cholesterol levels and the consumption of stanol ester enriched liquid yoghurt. The alternative hypothesis establishes a relationship between such consumption and the incidence of the primary variable.

The main objective of this study is to determine the efficacy of the intake of 2 g of plant sterol esters a day in lowering LDL-cholesterol levels in patients diagnosed with hypercholesterolaemia. The specific objectives are: 1) to quantify the efficacy of the daily intake of plant sterol esters in lowering LDL-cholesterol, total cholesterol and cardiovascular risk in patients with hypercholesterolaemia; 2) to evaluate the occurrence of adverse effects of the daily intake of plant sterol esters; 3) to identify the factors that determine a greater reduction in lipid levels in subjects receiving plant sterol ester supplements.

Study design Randomised, double-blind, placebo controlled experimental trial carried out at family doctors' surgeries at three health centres in the Health Area of Albacete (Spain). The study subjects will be adults diagnosed with "limit" or "defined" hypercholesterolaemia and who have LDL cholesterol levels of 130 mg/dl or over. A dairy product in the form of liquid yoghurt containing 2 g of plant sterol ester per container will be administered daily after the main meal, for a period of 24 months. The control group will receive a daily unit of yogurt not supplemented with plant sterol esters that has a similar appearance to the enriched yoghurt. The primary variable is the change in lipid profile at 1, 3, 6, 12, 18 and 24 months. The secondary variables are: change in cardiovascular risk, adherence to the dairy product, adverse effects, adherence to dietary recommendations, frequency of food consumption, basic physical examination data, health problems, lipid-lowering medication, physical activity, smoking habits and socio-demographic variables.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with limit hypercholesterolaemia (total cholesterol 200-249 mg/dl) or defined hypercholesterolaemia (total cholesterol equal to or above 250 mg/dl) who have LDL-cholesterol levels equal to or above 130 mg/dl
* Subjects aged 18 years or over attending the participating health centres
* Subjects who give their consent to participate after being informed of the study objectives

Exclusion Criteria:

* Known hypersensitivity to sterol esters or to the other components of the food that contains them (liquid yoghurt)
* Contraindication for treatment with sterol esters or any of the components of the food
* Physical disability that hinders collaboration
* Significant chronic organic or psychiatric disease
* Not obtaining informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change in lipid profile | At 1, 3, 6, 12, 18 and 24 months
  Lipid levels will be measured in both plasma and capillary blood at the initial visit. The validity of the capillary blood lipid levels can be checked with the Cardiochek analyser (by total cholesterol, HDL-cholesterol and triglyceride strips, and subsequent calculation of LDL-cholesterol using the Friedewald formula). The measurements at 3, 12 and 24 months will be in plasma. At 1, 6 and 18 months they will only be in capillary blood.

SECONDARY OUTCOMES:
Change in cardiovascular risk | At 1, 3, 6, 12, 18 and 24 months
  SCORE and REGICOR tables will be used for the evaluation.
Adherence to the dairy product (liquid yoghurt) | At 1, 3, 6, 12, 18 and 24 months
  By self-report and Morisky-Green scale, which determines the degree of coincidence between the patient's behaviour and the doctor's advice (a non-complier is one who answers one of the four questions of the scale inappropriately).
Adverse events | At 1, 3, 6, 12, 18 and 24 months
  Considered as any undesirable event in any patient included in the study, even though it does not have a causal relation with the product. Known adverse events of phytosterols in the diet at the proposed doses: occasionally mild digestive alterations.
Adherence to the dietary recommendations | At 1, 3, 6, 12, 18 and 24 months
  5-point Likert scale
Frequency of food intake | At 1, 3, 6, 12, 18 and 24 months
  Using the CDC-FFQ questionnaire, validated in Spain (Aguirre, 2008) considered appropriate to classify the subjects according to their intake of food and nutrients.
Occurrence of cardiovascular events | At 1, 3, 6, 12, 18 and 24 months
  Ischaemic heart disease, atherothrombotic cerebrovascular disease, heart failure and peripheral artery disease.
  -Weight, height, body mass index (BMI): classification of subjects according to degree of obesity.
Weight, height, body mass index (BMI) | At 1, 3, 6, 12, 18 and 24 months
  Classification of subjects according to degree of obesity.
Physical activity | At 1, 3, 6, 12, 18 and 24 months
  Amount of aerobic exercise ("active" if performs aerobic exercise for 30 minutes or more, three or more times a week, "partially active" if exercises with less frequency and for less time that this and "inactive" when does not perform any type of exercise).
Smoking habit | At 1, 3, 6, 12, 18 and 24 months
  Considered smoker if answers yes to the question "do you smoke?"
Systolic and diastolic blood pressure (two measurements): | At 1, 3, 6, 12, 18 and 24 months
  The result will be the mean of the two measurements.
Health problems | At 1, 3, 6, 12, 18 and 24 months
  (WONCA ICPC-2)
Lipid-lowering pharmacological treatment. | At 1, 3, 6, 12, 18 and 24 months
  Whether taking lipid-lowering pharmacological treatment.
Socio-demographic data | Initial visit
  Age, gender, marital status, educational level and social class based on occupation (National Classification of Occupations).

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Párraga, PhD, Principal Investigator — Research Unit. Primary Care Head Office of Albacete; Jesús López-Torres, PhD, Study Chair — Research Unit. Primary Care Head Office of Albacete.; Fernando Andrés, Bachelor of Computer Sciences, Study Chair — Research Unit. Primary Care Head Office of Albacete.; Beatriz Navarro, PhD, Study Chair — Research Unit. Primary Care Head Office of Albacete.; José María Del Campo, PhD, Study Chair — Primary Care Head Office of Albacete.; Mercedes García-Reyes, PhD, Study Chair — Primary Care Head Office of Albacete.; María Pilar Galdón, PhD, Study Chair — Primary Care Head Office of Albacete.; Ángeles Lloret, Bachelor of Pharmacy, Study Chair — Primary Care Head Office of Albacete.; Juan Carlos Precioso, Bachelor of Medicine, Study Chair — Primary Care Head Office of Albacete.; Joseba Rabanales, Bachelor of Nursing, Study Chair — Research Unit. Primary Care Head Office of Albacete.

REFERENCES:
- [Background] Medrano MJ, Cerrato E, Boix R, Delgado-Rodriguez M. [Cardiovascular risk factors in Spanish population: metaanalysis of cross-sectional studies]. Med Clin (Barc). 2005 Apr 30;124(16):606-12. doi: 10.1157/13074389. Spanish. PMID 15871776
- [Background] Gutierrez Fuentes JA, Gomez-Jerique J, Gomez De La Camara A, Angel Rubio M, Garcia Hernandez A, Aristegui I; Diet and Cardiovascular Risk in Spain Study (DRECE II). [Diet and cardiovascular risk in Spain. Description of the evolution of cardiovascular prolile]. Med Clin (Barc). 2000 Dec 2;115(19):726-9. Spanish. PMID 11141438
- [Background] Law MR, Wald NJ, Thompson SG. By how much and how quickly does reduction in serum cholesterol concentration lower risk of ischaemic heart disease? BMJ. 1994 Feb 5;308(6925):367-72. doi: 10.1136/bmj.308.6925.367. PMID 8043072
- [Background] Law MR, Wald NJ. Risk factor thresholds: their existence under scrutiny. BMJ. 2002 Jun 29;324(7353):1570-6. doi: 10.1136/bmj.324.7353.1570. No abstract available. PMID 12089098
- [Background] Keys A. Coronary heart disease, serum cholesterol, and the diet. Acta Med Scand. 1980;207(3):153-60. doi: 10.1111/j.0954-6820.1980.tb09697.x. No abstract available. PMID 7368981
- [Background] Baigent C, Keech A, Kearney PM, Blackwell L, Buck G, Pollicino C, Kirby A, Sourjina T, Peto R, Collins R, Simes R; Cholesterol Treatment Trialists' (CTT) Collaborators. Efficacy and safety of cholesterol-lowering treatment: prospective meta-analysis of data from 90,056 participants in 14 randomised trials of statins. Lancet. 2005 Oct 8;366(9493):1267-78. doi: 10.1016/S0140-6736(05)67394-1. Epub 2005 Sep 27. PMID 16214597
- [Background] McCullough ML, Feskanich D, Stampfer MJ, Giovannucci EL, Rimm EB, Hu FB, Spiegelman D, Hunter DJ, Colditz GA, Willett WC. Diet quality and major chronic disease risk in men and women: moving toward improved dietary guidance. Am J Clin Nutr. 2002 Dec;76(6):1261-71. doi: 10.1093/ajcn/76.6.1261. PMID 12450892
- [Background] Sudhop T, von Bergmann K. Cholesterol absorption inhibitors for the treatment of hypercholesterolaemia. Drugs. 2002;62(16):2333-47. doi: 10.2165/00003495-200262160-00002. PMID 12396226
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner DA, Wong JM, de Souza R, Emam A, Parker TL, Vidgen E, Trautwein EA, Lapsley KG, Josse RG, Leiter LA, Singer W, Connelly PW. Direct comparison of a dietary portfolio of cholesterol-lowering foods with a statin in hypercholesterolemic participants. Am J Clin Nutr. 2005 Feb;81(2):380-7. doi: 10.1093/ajcn.81.2.380. PMID 15699225
- [Background] Bellisle F, Blundell JE, Dye L, Fantino M, Fern E, Fletcher RJ, Lambert J, Roberfroid M, Specter S, Westenhofer J, Westerterp-Plantenga MS. Functional food science and behaviour and psychological functions. Br J Nutr. 1998 Aug;80 Suppl 1:S173-93. doi: 10.1079/bjn19980109. PMID 9849358
- [Background] Ros E. [Introduction to functional food]. Med Clin (Barc). 2001 May 5;116(16):617-9. doi: 10.1016/s0025-7753(01)71924-0. No abstract available. Spanish. PMID 11412648
- [Background] Silveira Rodriguez MB, Monereo Megias S, Molina Baena B. [Functional nutrition and optimal nutrition. Near or far?]. Rev Esp Salud Publica. 2003 May-Jun;77(3):317-31. Spanish. PMID 12852326
- [Background] Cater NB. Plant stanol ester: review of cholesterol-lowering efficacy and implications for coronary heart disease risk reduction. Prev Cardiol. 2000 Summer;3(3):121-130. doi: 10.1111/j.1520-037x.2000.80370.x. PMID 11834929
- [Background] Hallikainen MA, Sarkkinen ES, Uusitupa MI. Plant stanol esters affect serum cholesterol concentrations of hypercholesterolemic men and women in a dose-dependent manner. J Nutr. 2000 Apr;130(4):767-76. doi: 10.1093/jn/130.4.767. PMID 10736328
- [Background] Miettinen TA, Puska P, Gylling H, Vanhanen H, Vartiainen E. Reduction of serum cholesterol with sitostanol-ester margarine in a mildly hypercholesterolemic population. N Engl J Med. 1995 Nov 16;333(20):1308-12. doi: 10.1056/NEJM199511163332002. PMID 7566021
- [Background] Miettinen TA, Vuoristo M, Nissinen M, Jarvinen HJ, Gylling H. Serum, biliary, and fecal cholesterol and plant sterols in colectomized patients before and during consumption of stanol ester margarine. Am J Clin Nutr. 2000 May;71(5):1095-102. doi: 10.1093/ajcn/71.5.1095. PMID 10799370
- [Background] Noakes M, Clifton PM, Doornbos AM, Trautwein EA. Plant sterol ester-enriched milk and yoghurt effectively reduce serum cholesterol in modestly hypercholesterolemic subjects. Eur J Nutr. 2005 Jun;44(4):214-22. doi: 10.1007/s00394-004-0513-z. Epub 2004 Aug 17. PMID 15316827
- [Background] Blair SN, Capuzzi DM, Gottlieb SO, Nguyen T, Morgan JM, Cater NB. Incremental reduction of serum total cholesterol and low-density lipoprotein cholesterol with the addition of plant stanol ester-containing spread to statin therapy. Am J Cardiol. 2000 Jul 1;86(1):46-52. doi: 10.1016/s0002-9149(00)00976-0. PMID 10867091
- [Background] Nigon F, Serfaty-Lacrosniere C, Beucler I, Chauvois D, Neveu C, Giral P, Chapman MJ, Bruckert E. Plant sterol-enriched margarine lowers plasma LDL in hyperlipidemic subjects with low cholesterol intake: effect of fibrate treatment. Clin Chem Lab Med. 2001 Jul;39(7):634-40. doi: 10.1515/CCLM.2001.103. PMID 11522112
- [Background] Gylling H, Miettinen TA. Combination therapy with statins. Curr Opin Investig Drugs. 2002 Sep;3(9):1318-23. PMID 12498007
- [Background] Katan MB, Grundy SM, Jones P, Law M, Miettinen T, Paoletti R; Stresa Workshop Participants. Efficacy and safety of plant stanols and sterols in the management of blood cholesterol levels. Mayo Clin Proc. 2003 Aug;78(8):965-78. doi: 10.4065/78.8.965. PMID 12911045
- [Background] Law M. Plant sterol and stanol margarines and health. BMJ. 2000 Mar 25;320(7238):861-4. doi: 10.1136/bmj.320.7238.861. No abstract available. PMID 10731187
- [Background] Mensink RP, Ebbing S, Lindhout M, Plat J, van Heugten MM. Effects of plant stanol esters supplied in low-fat yoghurt on serum lipids and lipoproteins, non-cholesterol sterols and fat soluble antioxidant concentrations. Atherosclerosis. 2002 Jan;160(1):205-13. doi: 10.1016/s0021-9150(01)00562-7. PMID 11755939
- [Background] O'Neill FH, Brynes A, Mandeno R, Rendell N, Taylor G, Seed M, Thompson GR. Comparison of the effects of dietary plant sterol and stanol esters on lipid metabolism. Nutr Metab Cardiovasc Dis. 2004 Jun;14(3):133-42. doi: 10.1016/s0939-4753(04)80033-4. PMID 15330272
- [Background] Mattson FH, Grundy SM, Crouse JR. Optimizing the effect of plant sterols on cholesterol absorption in man. Am J Clin Nutr. 1982 Apr;35(4):697-700. doi: 10.1093/ajcn/35.4.697. PMID 7072622
- [Background] Plat J, van Onselen EN, van Heugten MM, Mensink RP. Effects on serum lipids, lipoproteins and fat soluble antioxidant concentrations of consumption frequency of margarines and shortenings enriched with plant stanol esters. Eur J Clin Nutr. 2000 Sep;54(9):671-7. doi: 10.1038/sj.ejcn.1601071. PMID 11002377
- [Background] Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults. Executive Summary of The Third Report of The National Cholesterol Education Program (NCEP) Expert Panel on Detection, Evaluation, And Treatment of High Blood Cholesterol In Adults (Adult Treatment Panel III). JAMA. 2001 May 16;285(19):2486-97. doi: 10.1001/jama.285.19.2486. No abstract available. PMID 11368702
- [Background] Van Horn L, Ernst N. A summary of the science supporting the new National Cholesterol Education Program dietary recommendations: what dietitians should know. J Am Diet Assoc. 2001 Oct;101(10):1148-54. doi: 10.1016/s0002-8223(01)00283-8. No abstract available. PMID 11678485
- [Background] Lichtenstein AH, Deckelbaum RJ. AHA Science Advisory. Stanol/sterol ester-containing foods and blood cholesterol levels. A statement for healthcare professionals from the Nutrition Committee of the Council on Nutrition, Physical Activity, and Metabolism of the American Heart Association. Circulation. 2001 Feb 27;103(8):1177-9. doi: 10.1161/01.cir.103.8.1177. PMID 11222485
- [Background] American Heart Association Nutrition Committee; Lichtenstein AH, Appel LJ, Brands M, Carnethon M, Daniels S, Franch HA, Franklin B, Kris-Etherton P, Harris WS, Howard B, Karanja N, Lefevre M, Rudel L, Sacks F, Van Horn L, Winston M, Wylie-Rosett J. Diet and lifestyle recommendations revision 2006: a scientific statement from the American Heart Association Nutrition Committee. Circulation. 2006 Jul 4;114(1):82-96. doi: 10.1161/CIRCULATIONAHA.106.176158. Epub 2006 Jun 19. PMID 16785338
- [Background] Algorta Pineda J, Chinchetru Ranedo MJ, Aguirre Anda J, Francisco Terreros S. [Hypocholesteremic effectiveness of a yogurt containing plant stanol esters]. Rev Clin Esp. 2005 Feb;205(2):63-6. doi: 10.1157/13072497. Spanish. PMID 15766477
- [Background] Slesinski RS, Turnbull D, Frankos VH, Wolterbeek AP, Waalkens-Berendsen DH. Developmental toxicity study of vegetable oil-derived stanol fatty acid esters. Regul Toxicol Pharmacol. 1999 Apr;29(2 Pt 1):227-33. doi: 10.1006/rtph.1999.1292. PMID 10341155
- [Background] De Jong N, Pijpers L, Bleeker JK, Ocke MC. Potential intake of phytosterols/-stanols: results of a simulation study. Eur J Clin Nutr. 2004 Jun;58(6):907-19. doi: 10.1038/sj.ejcn.1601912. PMID 15164112
- [Background] Brufau G, Canela MA, Rafecas M. Phytosterols: physiologic and metabolic aspects related to cholesterol-lowering properties. Nutr Res. 2008 Apr;28(4):217-25. doi: 10.1016/j.nutres.2008.02.003. PMID 19083411
- [Background] Moruisi KG, Oosthuizen W, Opperman AM. Phytosterols/stanols lower cholesterol concentrations in familial hypercholesterolemic subjects: a systematic review with meta-analysis. J Am Coll Nutr. 2006 Feb;25(1):41-8. doi: 10.1080/07315724.2006.10719513. PMID 16522931
- [Background] Jordan S, Griffiths J, Pilon K. Sterol and sterolin-containing products: hematologic adverse reactions. CMAJ. 2004 Apr 13;170(8):1347-8, 1351-2. No abstract available. English, French. PMID 15108714
- [Background] Hallikainen MA, Sarkkinen ES, Uusitupa MI. Effects of low-fat stanol ester enriched margarines on concentrations of serum carotenoids in subjects with elevated serum cholesterol concentrations. Eur J Clin Nutr. 1999 Dec;53(12):966-9. doi: 10.1038/sj.ejcn.1600882. PMID 10602355
- [Background] Noakes M, Clifton P, Ntanios F, Shrapnel W, Record I, McInerney J. An increase in dietary carotenoids when consuming plant sterols or stanols is effective in maintaining plasma carotenoid concentrations. Am J Clin Nutr. 2002 Jan;75(1):79-86. doi: 10.1093/ajcn/75.1.79. PMID 11756063
- [Background] Rajaratnam RA, Gylling H, Miettinen TA. Independent association of serum squalene and noncholesterol sterols with coronary artery disease in postmenopausal women. J Am Coll Cardiol. 2000 Apr;35(5):1185-91. doi: 10.1016/s0735-1097(00)00527-1. PMID 10758959
- [Background] Assmann G, Cullen P, Erbey J, Ramey DR, Kannenberg F, Schulte H. Plasma sitosterol elevations are associated with an increased incidence of coronary events in men: results of a nested case-control analysis of the Prospective Cardiovascular Munster (PROCAM) study. Nutr Metab Cardiovasc Dis. 2006 Jan;16(1):13-21. doi: 10.1016/j.numecd.2005.04.001. Epub 2005 Jul 28. PMID 16399487
- [Background] Moghadasian MH, McManus BM, Godin DV, Rodrigues B, Frohlich JJ. Proatherogenic and antiatherogenic effects of probucol and phytosterols in apolipoprotein E-deficient mice: possible mechanisms of action. Circulation. 1999 Apr 6;99(13):1733-9. doi: 10.1161/01.cir.99.13.1733. PMID 10190884
- [Background] Volger OL, Mensink RP, Plat J, Hornstra G, Havekes LM, Princen HM. Dietary vegetable oil and wood derived plant stanol esters reduce atherosclerotic lesion size and severity in apoE*3-Leiden transgenic mice. Atherosclerosis. 2001 Aug;157(2):375-81. doi: 10.1016/s0021-9150(00)00750-4. PMID 11472737
- [Background] Ratnayake WM, L'Abbe MR, Mueller R, Hayward S, Plouffe L, Hollywood R, Trick K. Vegetable oils high in phytosterols make erythrocytes less deformable and shorten the life span of stroke-prone spontaneously hypertensive rats. J Nutr. 2000 May;130(5):1166-78. doi: 10.1093/jn/130.5.1166. PMID 10801914
- [Background] Child P, Kuksis A. Differential uptake of cholesterol and plant sterols by rat erythrocytes in vitro. Lipids. 1982 Oct;17(10):748-54. doi: 10.1007/BF02534662. PMID 7176832
- [Background] de Jong A, Plat J, Mensink RP. Plant sterol or stanol consumption does not affect erythrocyte osmotic fragility in patients on statin treatment. Eur J Clin Nutr. 2006 Aug;60(8):985-90. doi: 10.1038/sj.ejcn.1602409. Epub 2006 Feb 15. PMID 16482072
- [Background] Hendriks HF, Brink EJ, Meijer GW, Princen HM, Ntanios FY. Safety of long-term consumption of plant sterol esters-enriched spread. Eur J Clin Nutr. 2003 May;57(5):681-92. doi: 10.1038/sj.ejcn.1601598. PMID 12771969
- [Derived] Parraga-Martinez I, Lopez-Torres-Hidalgo JD, Del Campo-Del Campo JM, Galdon-Blesa MP, Precioso-Yanez JC, Rabanales-Sotos J, Garcia-Reyes-Ramos M, Andres-Pretel F, Navarro-Bravo B, Lloret-Callejo A. Long-term Effects of Plant Stanols on the Lipid Profile of Patients With Hypercholesterolemia. A Randomized Clinical Trial. Rev Esp Cardiol (Engl Ed). 2015 Aug;68(8):665-71. doi: 10.1016/j.rec.2014.07.035. Epub 2014 Dec 23. PMID 25541227
- [Derived] Parraga I, Lopez-Torres J, Andres F, Navarro B, del Campo JM, Garcia-Reyes M, Galdon MP, Lloret A, Precioso JC, Rabanales J. Effect of plant sterols on the lipid profile of patients with hypercholesterolaemia. Randomised, experimental study. BMC Complement Altern Med. 2011 Sep 12;11:73. doi: 10.1186/1472-6882-11-73. PMID 21910898